CLINICAL TRIAL: NCT04796987
Title: Convolutional Neural Network for the Detection of Cervical Myelomalacia on Magnetic Resonance Imaging
Brief Title: Convolutional Neural Network for the Detection of Cervical Myelomalacia
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Principle investigator, Istanbul University
Other Study IDs: KAEK/2020.07.129
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Cervical Myelopathy
Keywords: neural network; deep learning; cervical myelopathy
MeSH Terms: interventions — Convolutional Neural Networks

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cervical myelopathy: MR images of patients with cervical myelopathy
  Interventions: Diagnostic Test: Convolutional Neural Network
- normal: normal section of the MRI of patients with cervical myelopathy
  Interventions: Diagnostic Test: Convolutional Neural Network

INTERVENTIONS:
Diagnostic Test: Convolutional Neural Network — Convolutional neural networks, a machine learning technique, have been used in several industrial and research fields increasingly. The development of computational units and the increasing amount of data led to the development of new methods on artificial neural networks. Deep learning (DL) is a multi-layered neural network in which feature extraction is done automatically. It extends traditional neural networks by adding more hidden layers to the network architecture between the input and output layers to model more complex and nonlinear relationships.

SUMMARY:
Deep learning technology has been used increasingly in spine surgery as well as in many medical fields. However, it is noticed that most of the studies about this subject in the literature have been conducted except of the cervical spine. In this study, we aimed to demonstrate the effectiveness of the deep learning algorithm in the diagnosis of cervical myelomalacia compared to conventional diagnostic methods.

Artificial neural networks, a machine learning technique, have been used in several industrial and research fields increasingly. The development of computational units and the increasing amount of data led to the development of new methods on artificial neural networks

DETAILED DESCRIPTION:
Cervical myelopathy (CM) is a frequent degenerative disease of the cervical spine that occurs as a result of compression of the spinal cord. In evaluating of this disease and determining treatment options, the patient's clinic and radiological modalities should be evaluated together.

The current imaging procedures for CM are plain roentgenograms, computed tomography and magnetic resonance imaging (MRI). However, MRI in CM is more valuable in evaluating of the disc, spinal cord and other soft tissues compared to other imaging methods. Artificial intelligence technologies also used in many health applications such as medical image analysis, biological signal analysis, etc. In this study, we aimed to demonstrate the effectiveness of the deep learning algorithm in the diagnosis of cervical myelomalacia compared to conventional diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

* the patients with classical cervical myelomalacia sypmtoms such as neck pain and stiffness, weakness and clumsiness at the upper extremities or gait difficulties and radiological findings of spinal compression
* 30-80 years age.

Exclusion Criteria:

* Patients with a previous history of cervical spinal surgery and has a systematic disease (rheumatologic or neural disease) .

Ages: 32 Years to 77 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants are aged 30-80 years, who have cervical myelomalacia that proved in MRI.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
The value of confusion matrix accuracy for sagittal views | 1 day
  It is a specific table layout that allows visualization of the performance of an algorithm.
The value of confusion matrix accuracy for axial views | 1 day
  It is a specific table layout that allows visualization of the performance of an algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Yilmaz, Principal Investigator — Karabuk University, Faculty of Engineering; Murat Korkmaz, Principal Investigator — Istanbul University, Faculty of Medicine
Locations (1):
- İstanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It can be shared after publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after publication